CLINICAL TRIAL: NCT03543566
Title: Antimuscarinic Medication for Urgency Urinary Incontinence in Women With Dual Incontinence (Darifenacin for Treatment of Women With Dual Incontinence)
Brief Title: Bladder Antimuscarinic Medication and Accidental Bowel Leakage
Acronym: BAMA
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Lindsay M Kissane, MD, University of Alabama at Birmingham
Other Study IDs: IRB-300000103
Record Dates: First submitted 2018-03-20; First posted 2018-06-01 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Urinary Incontinence, Urge; Fecal Incontinence
Keywords: antimuscarinic medication; medical management; dual incontinence; darifenacin; quality of life; bowel diary
MeSH Terms: conditions — Urinary Incontinence, Urge; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational research study will examine whether a medication known as darifenacin (Enablex ®) used for urgency urinary incontinence (UUI) also helps to improve fecal incontinence symptoms. Darifenacin is FDA approved for UUI, but is not FDA approved for fecal incontinence or specifically for dual incontinence (treatment of urinary incontinence and fecal incontinence at the same time). If participants are eligible for this study, they will have had symptoms of bothersome urgency urinary incontinence and fecal incontinence, and have decided to try medication for urgency urinary incontinence. Darifenacin (Enablex ®) is an oral medication which relaxes the bladder muscle to help prevent urgency urinary leakage. It is commonly used to treat overactive bladder and urgency urinary leakage. There is some evidence that this medication may also help with fecal incontinence by slowing the gut and preventing loose stools. Investigators are planning to enroll approximately 30 patients who have both UUI and fecal incontinence and who choose medical treatment as a part of their standard care.

DETAILED DESCRIPTION:
Urgency urinary incontinence (UUI) and fecal incontinence (FI) are two highly prevalent pelvic floor disorders which negatively impact quality of life (QOL). Among women with urgency urinary incontinence (UUI), 8-20% also suffer from FI.

Initial management of both UUI and FI consists of behavioral therapies with or without pharmacologic management. First line management of FI includes diet, fluid and fiber intake adjustments (Grade A), antidiarrheal medication (Grade B) and exercises to strengthen and enhance awareness of the anal sphincter (Grade C). If symptoms fail to improve with these measures by 8-12 weeks, further investigations should be considered before moving to more invasive management options such as bulking agents, sphincterplasty or sacral nerve stimulation.

In addition to fiber and antidiarrheals, medications with antimuscarinic effects such as hyoscyamine and tricyclic antidepressants are often used in the treatment of FI and IBS-D. Antimuscarinic medications function in this setting by blockade of colonic muscarinic acetylcholine receptors causing smooth muscle relaxation, decreased gut motility and prolonged colon transit time.

In patients with overactive bladder (OAB) with UUI, anti-muscarinic medications or a β3-adrenoreceptor agonist medication can be added to behavioral therapy as first line to optimize symptom control and QOL (Gormley 2015). In patients being treated for UUI, constipation is often viewed as an unwanted side effect of antimuscarinic medications, with varying constipation rates observed among the different medications. Non-selective antimuscarinic medications such as fesoterodine (Toviaz ®) and tolterodine (Detrol ®) may be less likely to cause constipation, whereas newer M2 or M3-selective agents such as darifenacin (Enablex ®), solifencin (Vesicare®) or trospium (Sanctura ®) may be more constipating. Darifenacin is notable for the highest constipation rates- up to 15% for the 7.5mg dose, and up to 21% for the 15mg dose.

While there is no current evidence for one specific antimuscarinic medication use in patients suffering with dual incontinence (specifically UUI and FI), many providers use the more constipating antimuscarinic medications as treatment in this setting. Patients with loose-stool-predominant FI may benefit from the constipating side effects by slowed colonic transit time, firmer bowel movements and thereby improved bowel-related QOL. Only one study has previously examined the effect of antimuscarinic medication for OAB on bowel-related QOL. In this descriptive study, 90 patients who were treated with antimuscarinic medication for OAB were followed to measure change in ePAQ (electronic Personal Assessment Questionnaire) score. Investigators reported significant improvement in bowel-related QOL three to six months after treatment. Authors did not specify pre-treatment diagnoses, symptoms or details of the antimuscarinic treatment.

While anecdotally antimuscarinic medications are an effective first line medication in patients with dual incontinence, more evidence is needed. The goal of our study therefore, is to observe the effect of standard of care antimuscarinic therapy for UUI on fecal incontinence symptoms in women with dual incontinence. Investigators will compare patient reported fecal incontinence symptoms before and after treatment in women with dual incontinence who elect to undergo standard of care medical management for UUI with the antimuscarinic medication darifenacin.

Hypothesis: In patients with dual incontinence, treatment of urgency urinary incontinence with darifenacin 7.5mg will improve FI symptom severity at 8 weeks Primary Aim: To characterize change in FI symptom severity (change in Vaizey score) after darifenacin treatment in patients with dual incontinence at 8 weeks

Secondary Aims:

Secondary Aim #1: To characterize post-treatment change in FI frequency using 7-day bowel diaries, change in quality of life (change in Fecal Incontinence Quality of Life (FIQOL) total and subscale scores), and characterize treatment improvement using the Patient Global Impression of Improvement (PGI-I) measure Secondary Aim #2: To describe compliance and adverse effects of antimuscarinic medication in patients with dual incontinence.

Secondary Aim #3: To describe effect of antimuscarinic medication on OAB symptom bother and quality of life in patients with dual incontinence, using the OAB questionnaire short form (OAB-q SF)

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18yrs presenting to UAB urogynecology and continence clinics with co-occurring UUI and FI
* Willing to complete all study related items

Exclusion Criteria:

* Severe constipation, fecal impaction or overflow fecal incontinence
* Inflammatory bowel disease, colorectal CA, spinal cord injury, multiple sclerosis, stroke, myasthenia gravis
* Infectious diarrhea
* Bothersome SUI (defined as "moderately" or greater bother on UDI-3)
* Patients planning to undergo surgery during study period
* Patients who are pregnant or intending to become pregnant during the study period
* Patients with contraindications to antimuscarinic medications (ie. closed angle glaucoma)
* Patients on unstable or changing dosage of fiber or narcotics in the past 14 days
* Patients taking more than 2mg/day of loperamide (patients taking more than 2mg will be required a 2 week washout period)
* Patients currently taking medication for urgency urinary incontinence (these patients will also require a 2 week washout period)
* Patients initiating care with a pelvic floor physical therapist during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patients only
Study Population: patients presenting to UAB urogynecology and continence clinics
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
change in FI symptom severity | 8 weeks
  to be measured by questionnaire and bowel diary Questionnaire to be used is the Vaizey scale which measures fecal incontinence severity. Minimum score is 0 (perfect continence; best) and maximum score is 24 (total incontinence; worse). There is no subscale.
  Bowel diary is a weeklong record of each bowel movement the patient has. there is no standardized scoring or scale.

SECONDARY OUTCOMES:
post-treatment change in FI frequency | 8 weeks
  to be measured by bowel diary
  Bowel diary is a weeklong record of each bowel movement the patient has. there is no standardized scoring or scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Kissane, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan SA, Dmochowski R, Cash BD, Kopp ZS, Berriman SJ, Khullar V. Systematic review of the relationship between bladder and bowel function: implications for patient management. Int J Clin Pract. 2013 Mar;67(3):205-16. doi: 10.1111/ijcp.12028. PMID 23409689
- [Background] Khullar V, Damiano R, Toozs-Hobson P, Cardozo L. Prevalence of faecal incontinence among women with urinary incontinence. Br J Obstet Gynaecol. 1998 Nov;105(11):1211-3. doi: 10.1111/j.1471-0528.1998.tb09978.x. PMID 9853773
- [Background] Coyne KS, Cash B, Kopp Z, Gelhorn H, Milsom I, Berriman S, Vats V, Khullar V. The prevalence of chronic constipation and faecal incontinence among men and women with symptoms of overactive bladder. BJU Int. 2011 Jan;107(2):254-61. doi: 10.1111/j.1464-410X.2010.09446.x. PMID 20590548
- [Background] Lawrence JM, Lukacz ES, Nager CW, Hsu JW, Luber KM. Prevalence and co-occurrence of pelvic floor disorders in community-dwelling women. Obstet Gynecol. 2008 Mar;111(3):678-85. doi: 10.1097/AOG.0b013e3181660c1b. PMID 18310371
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Kannan H, Radican L, Turpin RS, Bolge SC. Burden of illness associated with lower urinary tract symptoms including overactive bladder/urinary incontinence. Urology. 2009 Jul;74(1):34-8. doi: 10.1016/j.urology.2008.12.077. Epub 2009 May 9. PMID 19428076
- [Background] Darkow T, Fontes CL, Williamson TE. Costs associated with the management of overactive bladder and related comorbidities. Pharmacotherapy. 2005 Apr;25(4):511-9. doi: 10.1592/phco.25.4.511.61033. PMID 15977912
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Brown HW, Wexner SD, Segall MM, Brezoczky KL, Lukacz ES. Quality of life impact in women with accidental bowel leakage. Int J Clin Pract. 2012 Nov;66(11):1109-16. doi: 10.1111/ijcp.12017. PMID 23067035
- [Background] Smith TM, Menees SB, Xu X, Saad RJ, Chey WD, Fenner DE. Factors associated with quality of life among women with fecal incontinence. Int Urogynecol J. 2013 Mar;24(3):493-9. doi: 10.1007/s00192-012-1889-6. Epub 2012 Jul 18. PMID 22806489
- [Background] Soligo M, Salvatore S, Milani R, Lalia M, Malberti S, Digesu GA, Mariani S. Double incontinence in urogynecologic practice: a new insight. Am J Obstet Gynecol. 2003 Aug;189(2):438-43. doi: 10.1067/s0002-9378(03)00466-6. PMID 14520214
- [Background] Lacima G, Espuna M, Pera M, Puig-Clota M, Quinto L, Garcia-Valdecasas JC. Clinical, urodynamic, and manometric findings in women with combined fecal and urinary incontinence. Neurourol Urodyn. 2002;21(5):464-9. doi: 10.1002/nau.10025. PMID 12232882
- [Background] Markland AD, Goode PS, Burgio KL, Redden DT, Richter HE, Sawyer P, Allman RM. Correlates of urinary, fecal, and dual incontinence in older African-American and white men and women. J Am Geriatr Soc. 2008 Feb;56(2):285-90. doi: 10.1111/j.1532-5415.2007.01509.x. Epub 2007 Dec 7. PMID 18070007
- [Background] Markland AD, Richter HE, Kenton KS, Wai C, Nager CW, Kraus SR, Xu Y, Tennstedt SL; Urinary Incontinence Treatment Network. Associated factors and the impact of fecal incontinence in women with urge urinary incontinence: from the Urinary Incontinence Treatment Network's Behavior Enhances Drug Reduction of Incontinence study. Am J Obstet Gynecol. 2009 Apr;200(4):424.e1-8. doi: 10.1016/j.ajog.2008.11.023. Epub 2009 Feb 6. PMID 19200939
- [Background] Whitehead WE, Borrud L, Goode PS, Meikle S, Mueller ER, Tuteja A, Weidner A, Weinstein M, Ye W; Pelvic Floor Disorders Network. Fecal incontinence in US adults: epidemiology and risk factors. Gastroenterology. 2009 Aug;137(2):512-7, 517.e1-2. doi: 10.1053/j.gastro.2009.04.054. Epub 2009 May 4. PMID 19410574
- [Background] Bharucha AE, Zinsmeister AR, Schleck CD, Melton LJ 3rd. Bowel disturbances are the most important risk factors for late onset fecal incontinence: a population-based case-control study in women. Gastroenterology. 2010 Nov;139(5):1559-66. doi: 10.1053/j.gastro.2010.07.056. Epub 2010 Aug 10. PMID 20708007
- [Background] Markland AD, Goode PS, Burgio KL, Redden DT, Richter HE, Sawyer P, Allman RM. Incidence and risk factors for fecal incontinence in black and white older adults: a population-based study. J Am Geriatr Soc. 2010 Jul;58(7):1341-6. doi: 10.1111/j.1532-5415.2010.02908.x. Epub 2010 Jun 1. PMID 20533967
- [Background] Freeman A, Menees S. Fecal Incontinence and Pelvic Floor Dysfunction in Women: A Review. Gastroenterol Clin North Am. 2016 Jun;45(2):217-37. doi: 10.1016/j.gtc.2016.02.002. PMID 27261895
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Background] Santoro GA, Eitan BZ, Pryde A, Bartolo DC. Open study of low-dose amitriptyline in the treatment of patients with idiopathic fecal incontinence. Dis Colon Rectum. 2000 Dec;43(12):1676-81; discussion 1681-2. doi: 10.1007/BF02236848. PMID 11156450
- [Background] Lucak S, Chang L, Halpert A, Harris LA. Current and emergent pharmacologic treatments for irritable bowel syndrome with diarrhea: evidence-based treatment in practice. Therap Adv Gastroenterol. 2017 Feb;10(2):253-275. doi: 10.1177/1756283X16663396. Epub 2016 Sep 16. PMID 28203283
- [Background] Ehrenpreis ED, Chang D, Eichenwald E. Pharmacotherapy for fecal incontinence: a review. Dis Colon Rectum. 2007 May;50(5):641-9. doi: 10.1007/s10350-006-0778-9. PMID 17205204
- [Background] Wang JY, Abbas MA. Current management of fecal incontinence. Perm J. 2013 Summer;17(3):65-73. doi: 10.7812/TPP/12-064. PMID 24355892
- [Background] Gormley EA, Lightner DJ, Burgio KL, Chai TC, Clemens JQ, Culkin DJ, Das AK, Foster HE Jr, Scarpero HM, Tessier CD, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline. J Urol. 2012 Dec;188(6 Suppl):2455-63. doi: 10.1016/j.juro.2012.09.079. Epub 2012 Oct 24. PMID 23098785
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Meek PD, Evang SD, Tadrous M, Roux-Lirange D, Triller DM, Gumustop B. Overactive bladder drugs and constipation: a meta-analysis of randomized, placebo-controlled trials. Dig Dis Sci. 2011 Jan;56(1):7-18. doi: 10.1007/s10620-010-1313-3. Epub 2010 Jul 2. PMID 20596778
- [Background] Chapple C, Steers W, Norton P, Millard R, Kralidis G, Glavind K, Abrams P. A pooled analysis of three phase III studies to investigate the efficacy, tolerability and safety of darifenacin, a muscarinic M3 selective receptor antagonist, in the treatment of overactive bladder. BJU Int. 2005 May;95(7):993-1001. doi: 10.1111/j.1464-410X.2005.05454.x. PMID 15839920
- [Background] Leroi AM. The role of sacral neuromodulation in double incontinence. Colorectal Dis. 2011 Mar;13 Suppl 2:15-8. doi: 10.1111/j.1463-1318.2010.02520.x. PMID 21284797
- [Background] Bulchandani S, Toozs-Hobson P, Parsons M, McCooty S, Perkins K, Latthe P. Effect of anticholinergics on the overactive bladder and bowel domain of the electronic personal assessment questionnaire (ePAQ). Int Urogynecol J. 2015 Apr;26(4):533-7. doi: 10.1007/s00192-014-2527-2. Epub 2014 Oct 17. PMID 25323310
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Bliss DZ, Savik K, Jung HJ, Whitebird R, Lowry A, Sheng X. Dietary fiber supplementation for fecal incontinence: a randomized clinical trial. Res Nurs Health. 2014 Oct;37(5):367-78. doi: 10.1002/nur.21616. Epub 2014 Aug 23. PMID 25155992
- [Background] Bols EM, Hendriks EJ, Deutekom M, Berghmans BC, Baeten CG, de Bie RA. Inconclusive psychometric properties of the Vaizey score in fecally incontinent patients: a prospective cohort study. Neurourol Urodyn. 2010 Mar;29(3):370-7. doi: 10.1002/nau.20758. PMID 19634170
- [Background] Jelovsek JE, Chen Z, Markland AD, Brubaker L, Dyer KY, Meikle S, Rahn DD, Siddiqui NY, Tuteja A, Barber MD. Minimum important differences for scales assessing symptom severity and quality of life in patients with fecal incontinence. Female Pelvic Med Reconstr Surg. 2014 Nov-Dec;20(6):342-8. doi: 10.1097/SPV.0000000000000078. PMID 25185630
- [Background] Markland AD, Burgio KL, Whitehead WE, Richter HE, Wilcox CM, Redden DT, Beasley TM, Goode PS. Loperamide Versus Psyllium Fiber for Treatment of Fecal Incontinence: The Fecal Incontinence Prescription (Rx) Management (FIRM) Randomized Clinical Trial. Dis Colon Rectum. 2015 Oct;58(10):983-93. doi: 10.1097/DCR.0000000000000442. PMID 26347971
- [Background] Markland AD, Richter HE, Burgio KL, Wheeler TL 2nd, Redden DT, Goode PS. Outcomes of combination treatment of fecal incontinence in women. Am J Obstet Gynecol. 2008 Dec;199(6):699.e1-7. doi: 10.1016/j.ajog.2008.08.035. PMID 19084101
- [Background] Devroede G, Giese C, Wexner SD, Mellgren A, Coller JA, Madoff RD, Hull T, Stromberg K, Iyer S; SNS Study Group. Quality of life is markedly improved in patients with fecal incontinence after sacral nerve stimulation. Female Pelvic Med Reconstr Surg. 2012 Mar-Apr;18(2):103-12. doi: 10.1097/SPV.0b013e3182486e60. PMID 22453321
- [Background] Eric Jelovsek J, Markland AD, Whitehead WE, Barber MD, Newman DK, Rogers RG, Dyer K, Visco A, Sung VW, Sutkin G, Meikle SF, Gantz MG; Pelvic Floor Disorders Network. Controlling anal incontinence in women by performing anal exercises with biofeedback or loperamide (CAPABLe) trial: Design and methods. Contemp Clin Trials. 2015 Sep;44:164-174. doi: 10.1016/j.cct.2015.08.009. Epub 2015 Aug 18. PMID 26291917
- [Derived] Kissane LM, Martin KD, Meyer I, Richter HE. Effect of darifenacin on fecal incontinence in women with double incontinence. Int Urogynecol J. 2021 Sep;32(9):2357-2363. doi: 10.1007/s00192-020-04369-3. Epub 2020 Jun 15. PMID 32542466